CLINICAL TRIAL: NCT00177489
Title: Coordinating Center for Multisite Intervention Trial for Diverse Caregivers
Brief Title: Coordinating Center for Caregiver Intervention Trial
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Richard Schulz, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG13305
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Family Caregivers; Dementia; Alzheimer Disease; Randomized Controlled Trial; Intervention Studies
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): The intervention addressed caregiver depression, burden, self-care, and social support and care recipient problem behaviors through 12 in-home and telephone sessions over 6 months.
  Interventions: Behavioral: multicomponent psychosocial intervention
- Control (Other): Caregivers in the control group received 2 brief "check-in" telphone calls during the 6 month intervention.
  Interventions: Other: Control arm

INTERVENTIONS:
Behavioral: multicomponent psychosocial intervention — The intervention addressed caregiver depression, burden, self-care, and social support and care recipient problem behaviors through 12 in-home and telephone sessions over 6 months.
  Arms: Treatment
Other: Control arm — Caregivers in the control group received 2 brief "check-in" telephone calls during the 6-month intervention.
  Arms: Control

SUMMARY:
The primary goal of this study is to test a single multi-component intervention among family caregivers of persons with Alzheimer's disease or related disorders. The overall objectives of study are to 1) identify and reduce modifiable risk factors among diverse family caregivers of patients with Alzheimer's Disease or a related disorder, 2) enhance the quality of care of the care recipients, and 3) enhance the well-being of the caregivers.

DETAILED DESCRIPTION:
The proposed Coordinating Center (CC) will work with five sites and staff from the National Institute on Aging (NIA) and the National Institute of Nursing Research (NINR) to implement a multi-site caregiver intervention trial. The overall objective of this research program is to refine and test a multicomponent psychosocial intervention to reduce burden and depression among family caregivers of persons with Alzheimer's Disease or a related disorder. This competing renewal will build upon results obtained from its parent multi-site feasibility study, Resources for Enhancing Alzheimer's Caregiver Health (REACH) funded by the NIA/NINR as a cooperative agreement (UO1-AG13305). In the study proposed here, five intervention sites (Birmingham, Memphis, Miami, Palo Alto, and Philadelphia) will recruit 600 (120 per site) caregiver-care recipient dyads consisting of equal numbers of African Americans/Blacks, Hispanics/Latinos, and Caucasians/Whites. Caregivers will be randomized to either an in-home multicomponent intervention condition or a standardized information-only control condition.

The Coordinating Center at the University of Pittsburgh will work with the intervention site investigators and the NIA/NINR to support the implementation of the intervention study at each site and to collect and analyze a common database across sites.

ELIGIBILITY:
Caregiver Inclusion/Exclusion Criteria:

* Inclusion Criteria:

  1. Age: 21 years or older
  2. Family member of the care recipient
  3. Must live with care recipient or share cooking facilities
  4. Must have a telephone that will enable use of CTIS (Computer Telephone Integration System) system
  5. Must plan to remain in the recruitment area for the duration of the intervention and follow-up
  6. Caregiver role for more than 6 months
  7. Must provide on average 4 hours of supervision or direct assistance per day for the care recipient
  8. Risk Screening Tool: must have a total score of at least 1 for questions 1-3, and a total of at least 2 for questions 4-9

Exclusion Criteria:

1. Non-English, non-Spanish speaking
2. Active treatment (chemotherapy, radiation therapy) for cancer
3. Imminent placement of care recipient into a nursing home or with another caregiver (within 6 months)
4. Involvement in another clinical trial for caregivers
5. Participant in REACH I study
6. SPMSQ:> or = 4 errors*

   * If the caregiver has been inconsistent with answers or repeated answers during the screening process, then the interviewer administers the Short Portable Mental Status Questionnaire (SPMSQ). If the caregiver missed 4 or more questions, he/she was excluded from the study.

Care Recipient Inclusion/Exclusion Criteria

Inclusion Criteria:

a. NINCDS (MD diagnosis) of dementia or cognitive impairment (raw score on MMSE of 23 or less)

Exclusion Criteria:

1. Non-English, non-Spanish speaking
2. History of Parkinson's Disease or a stroke with no reported decline in memory over the past year
3. Active treatment (chemotherapy, radiation therapy) for cancer
4. More than three acute medical hospitalizations in past year (other than psychiatric or Alzheimer's Disease related admission)
5. Schizophrenia (onset of delusions before age 45) or other severe mental illness
6. Dementia secondary to head trauma (probable)
7. Blindness or deafness if either disability prohibits them from completion of data collection or participation in the interventions
8. MMSE = 0 and Bedbound (confined to a bed or chair for >22 hours per day, for at least 4 of the past 7 days)
9. Planned nursing home admission in 6 months
10. Participant in REACH I study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2002-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
multivariate quality of life indicator- assessed caregiver burden, depressive symptoms, self-care, social support and patient problem behaviors. Assessed at six months post-randomization. | six months

SECONDARY OUTCOMES:
Caregiver clinical depression and patient institutional placement-six months post-randomization. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schulz, Ph.D., Principal Investigator — Professor of Psychiatry and Director, University Center for Social and Urban Research, University of Pittsburgh
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University and Veterans Affairs, Menlo Park, California
  - University of Miami at Miami, Center on Adult Development and Aging, Miami, Florida
  - Thomas Jefferson University at Philadelphia, Center for Applied Research on Aging and Health, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
There is no plan to make individual participant data available.

REFERENCES:
- [Result] Belle SH, Burgio L, Burns R, Coon D, Czaja SJ, Gallagher-Thompson D, Gitlin LN, Klinger J, Koepke KM, Lee CC, Martindale-Adams J, Nichols L, Schulz R, Stahl S, Stevens A, Winter L, Zhang S; Resources for Enhancing Alzheimer's Caregiver Health (REACH) II Investigators. Enhancing the quality of life of dementia caregivers from different ethnic or racial groups: a randomized, controlled trial. Ann Intern Med. 2006 Nov 21;145(10):727-38. doi: 10.7326/0003-4819-145-10-200611210-00005. PMID 17116917
- [Derived] Nichols LO, Martindale-Adams J, Burns R, Graney MJ, Zuber J. Typical and atypical dementia family caregivers: systematic and objective comparisons. Int J Aging Hum Dev. 2011;72(1):27-43. doi: 10.2190/AG.72.1.b. PMID 21391405
- [Derived] Elliott AF, Burgio LD, Decoster J. Enhancing caregiver health: findings from the resources for enhancing Alzheimer's caregiver health II intervention. J Am Geriatr Soc. 2010 Jan;58(1):30-7. doi: 10.1111/j.1532-5415.2009.02631.x. PMID 20122038
- See also: REACH II website- click here for more information about this study — http://www.edc.gsph.pitt.edu/reach2